CLINICAL TRIAL: NCT01065116
Title: Effectiveness and Treatment Adherence to Artemether/Lumefantrine Pre-packs Versus Blister Packs in the Treatment of Uncomplicated Malaria in Uganda
Brief Title: Artemether-Lumefantrine (AL) Unit Dose Pre-packs Versus Blister Packs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Malaria Consortium, Uganda (Other)
Collaborators: Ministry of Health, Uganda (Other Government); Makerere University (Other)
Responsible Party: Nankabirwa Joaniter, Makerere University Kampala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMDIS -Blisterpack
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-05

CONDITIONS: Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AL Blister-pack (Experimental)
  Interventions: Drug: AL Blister-packs with Instruction leaflets
- AL unit dose age specific pre-packs (Active Comparator)
  Interventions: Drug: AL unit dose age specific pre-packs

INTERVENTIONS:
Drug: AL Blister-packs with Instruction leaflets — AL Blister packs with instruction leaflets will be dispensed
  Other Names: Coartem Blister packs
  Arms: AL Blister-pack
Drug: AL unit dose age specific pre-packs — Age specific colour coded Unit dose pre-packs will be used
  Other Names: Coartem pre-packs
  Arms: AL unit dose age specific pre-packs

SUMMARY:
The purpose of this study is to determine if adherence and effectiveness of AL in the treatment of uncomplicated malaria in children aged under five years using blister packs with pictorial leaflets can be at levels comparable to those with unit dosed age specific pre-packs.

DETAILED DESCRIPTION:
Prompt and adequate treatment of clinical malaria episodes remains one of the key elements of malaria control and this partly depends on patients' compliance to treatment. Uganda adopted Artemether-Lumefantrine (AL) as first line treatment for uncomplicated malaria. This is available at the health facilities in form of 6 dose pre-packs with different doze strengths in different packages. However, concerns about the costs and stock-outs of these packages have been raised and alternative equally efficacious alternatives need to be determined in order to reduce these problems. This study will assess if AL blister-packs can act as alternatives to the unit dose age specific pre-packs in the public sector

ELIGIBILITY:
Inclusion Criteria:

* Reported history of fever within last 48 hours and or an axillary temperature greater than or equal to 37.50C.
* Weight between 5 kg and 25 kg
* Positive malaria smear results for P. falciparum
* No history of intake of AL in the preceding two weeks
* Able to tolerate oral therapy
* Caregiver has given written informed consent to participate in the study
* If they reside within the designated catchment area of the health facility

Exclusion Criteria:

* Features of life threatening illness including severe malaria

Ages: 4 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 920 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Adherence to Blister-packs versus unit dose pre-packs as measured by pill count and self report. | Day 3

SECONDARY OUTCOMES:
Parasitological cure rates | Day 28
Clinical cure rates | Days 3

CONTACTS AND LOCATIONS:
Overall Officials: Joaniter I Nankabirwa, MSc CEB, Principal Investigator — Makerere University Kampala
Locations (1):
- Mulanda Health centre IV, Tororo District, Uganda, Uganda